CLINICAL TRIAL: NCT01661114
Title: A Trial of Gemcitabine, Infusional 5-Fluorouracil and Cisplatin for Advanced Pancreatic and Biliary Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2011.036; HUM 49518 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2012-07-24; First posted 2012-08-09 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-09

CONDITIONS: Pancreatic Cancer; Biliary Cancer
Keywords: Gemcitabine, Infusional 5-Fluorouracil,Cisplatin; Advanced Pancreatic and Biliary Cancers; untreated & previously treated pancreatic & biliary cancer.
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms | interventions — Gemcitabine; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, 5-FU and Cisplatin (Experimental): 4 cycles - Gemcitabine, 5-FU and Cisplatin (2 months)-Continue treatment until progression of disease or intolerable toxicity
  Interventions: Drug: Gemcitabine; Drug: 5-FU; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine
Drug: 5-FU
  Other Names: 5-Fluorouracil
Drug: Cisplatin

SUMMARY:
Multi-agent chemotherapy has value for patients with advanced pancreatic-biliary cancers leading to responses in a substantial minority and increasing survival. The use of the FOLFIRINOX regimen is limited by its' intensity and toxicity. Previous protocol and clinical experience within the University of Michigan Pancreatic Program leads to an expectation of tolerance and efficacy of the proposed regimen. Advantages of the proposed regimen relative to FOLFIRINOX include:

1. Substitution of gemcitabine for irinotecan. Single agent activity of gemcitabine is at least as good as irinotecan (probably better, especially when delivered by FDR [fixed-dose rate] infusion) and gemcitabine is much better tolerated with less diarrhea, nausea/emesis, myelosuppression and alopecia.
2. Deletion of leucovorin infusion and 5FU bolus injection will lessen myelosuppression, mucositis and diarrhea.
3. Substitution of cisplatin for oxaliplatin will reduce cost of therapy and avoid cold aggravated dysesthesia.

Presuming evidence of efficacy and confirmation of tolerance with the proposed regimen, the investigators believe this treatment may be more widely applicable to pancreatic-biliary cancer patients, including those with advanced disease as well as being considered for use in locally advanced and neo- and adjuvant settings.

DETAILED DESCRIPTION:
Gemcitabine combined with 5FU may enhance the activity of 5-FU in vivo. Gemcitabine is an inhibitor of ribonucleotide reductase, an enzyme needed for synthesis of deoxynucleotides, and 5-FU interferes with dTTP synthesis by inhibition of thymidylate synthase (TS). It is likely that concomitant administration of gemcitabine and 5FU results in increased cytotoxicity by reducing intracellular dTTP thru two different mechanisms, thereby inhibiting DNA replication and repair. Platinum compounds lead to cell death by forming DNA adducts and causing double strand breaks. By inhibiting DNA synthesis and repair, both gemcitabine and 5-FU potentiate the activity of cisplatin. These interactions underlie the clinical synergism that has been observed with platinum/5FU and platinum/gemcitabine combinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic or cytologic diagnosis of pancreatic adenocarcinoma or biliary tract cancer (intrahepatic or extrahepatic cholangiocarcinoma or gallbladder carcinoma).
* Patients must have clinical/radiologic evidence of metastatic disease.
* Previous systemic therapy for metastatic disease limited to one cytotoxic chemotherapy regimen not containing cisplatin. Previous therapy for metastatic disease might have included gemcitabine or infusional 5-FU but not both agents.
* ECOG (Eastern Cooperative Oncology Group) performance status < 1 (A measure of quality of life where 0 represents asymptomatic and 5 represents death).
* Patients must have adequate bone marrow (absolute neutrophil count >1,500/mm3, platelet count >100,000/mm3) and renal function (serum creatinine < 1.25 x ULN).
* Patients must have at least one measurable lesion per RECIST criteria.
* Patients must be free of serious concomitant medical disorders incompatible with study participation including active infection requiring systemic therapy.
* Previous malignancies are permitted provided that they have been treated with curative intent and patient is without evidence of active systemic disease.
* Patients must be informed of the investigational nature of this study and provide written informed consent prior to receiving protocol treatment.

Exclusion Criteria:

* Patients with pre-existing peripheral neuropathy > grade 2 are ineligible.
* Previous systemic therapy for metastatic disease limited to one cytotoxic chemotherapy regimen not containing cisplatin.
* Previous therapy for metastatic disease might have included gemcitabine or infusional 5-FU but not both agents.
* Serious concomitant medical disorders incompatible with study participation including active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Colucci et al., 2002, Louvet et al., 2005, Berlin et al., 2002, Cunningham et al., 2009, Heinemann et al., 2008, Valle et al., 2010

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine, 5-FU and Cisplatin
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, 5-FU and Cisplatin
Number analyzed (Participants) | 39
Age, Continuous [Mean (Full Range); unit: years] | 61 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Untreated and Previously Treated Patients That Had a Partial Response to Treatment
Description: The primary objective of this clinical trial is to estimate the response rate to treatment with the triplet chemotherapy regimen of gemcitabine, infusional 5-FU, and cisplatin, in untreated and previously treated advanced pancreatic and biliary cancer patients.
  Partial Response (PR) is defined as At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 28 days
Population: Patients with metastatic adenocarcinoma of the pancreas or biliary tract, previously untreated or having received one cytotoxic regimen for advanced disease.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Gemcitabine, 5-FU and Cisplatin
Number analyzed (Participants) | 39
percentage of patients
  Untreated | 40 [21.1 to 61.3]
  Received Previous Treatment | 7.1 [1.8 to 33.9]

2. Secondary Outcome: Median Overall Survival of Previously Treated and Previously Untreated Patients
Description: To assess the overall survival following treatment with gemcitabine, 5-FU and cisplatin.
Time Frame: 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine, 5-FU and Cisplatin
Number analyzed (Participants) | 39
Months
  Previously Untreated | 10.3 [8 to 19.4]
  Previously Treated | 4.9 [3.6 to 11.9]

ADVERSE EVENTS:
Arm/Group | Gemcitabine, 5-FU and Cisplatin
Serious Adverse Events (participants affected / at risk) | 10/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, 5-FU and Cisplatin (N=39)
Anal Ulcer (Gastrointestinal disorders) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 2 (2)
Joint infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, 5-FU and Cisplatin (N=39)
Anemia (Blood and lymphatic system disorders) | 36 (49)
Palpitations (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 3 (3)
Eye pain (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (9)
Anal ulcer (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (14)
Diarrhea (Gastrointestinal disorders) | 13 (18)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Duodenal obstruction (Gastrointestinal disorders) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 24 (38)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 15 (23)
Chills (General disorders) | 3 (4)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 4 (4)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 26 (36)
Fever (General disorders) | 9 (10)
Flu like symptoms (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Neck edema (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (4)
Pain (General disorders) | 4 (4)
Appendicitis (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 2 (2)
Joint infection (Infections and infestations) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 4 (5)
Urinary tract infection (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (12)
Alkaline phosphatase increased (Investigations) | 10 (12)
Aspartate aminotransferase increased (Investigations) | 8 (11)
Blood bilirubin increased (Investigations) | 6 (10)
Creatinine increased (Investigations) | 5 (6)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 29 (44)
Neutrophil count decreased (Investigations) | 27 (50)
Platelet count decreased (Investigations) | 29 (53)
Serum amylase increased (Investigations) | 1 (1)
Weight gain (Investigations) | 2 (3)
Weight loss (Investigations) | 11 (14)
White blood cell decreased (Investigations) | 31 (65)
Anorexia (Metabolism and nutrition disorders) | 13 (14)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 21 (29)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 13 (18)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 7 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 15 (19)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 6 (6)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (9)
Syncope (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (9)
Depression (Psychiatric disorders) | 4 (4)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (5)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes